CLINICAL TRIAL: NCT01861834
Title: A Safer Approach to Total Parenteral Nutrition in Pediatric Short Bowel Syndrome Intended to Decrease the Frequency and Severity of Liver Damage
Brief Title: Safer Parenteral Nutrition in Pediatric Short Bowel Syndrome to Decrease Liver Damage
Status: Approved for marketing | Type: Expanded Access
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: IND107300
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Cholestasis of Parenteral Nutrition
Keywords: Total parenteral nutrition; TPN; Intestinal Failure; Short Bowel Syndrome; Cholestasis; Intestinal failure associated liver disease; Parenteral nutrition associated liver disease
MeSH Terms: conditions — Hyperphagia; Intestinal Failure; Short Bowel Syndrome; Cholestasis

INTERVENTIONS:
Drug: Omegaven 10% — Patients with a sustained TPN requirement due to short bowel syndrome and TPN-associated liver disease that threatens progression to liver failure and death, for which the only available means of prevention at present is timely liver and/or intestinal transplant.
  Omegaven 10%, 1 gram/kg, IV, every 12 hours until transplantation, or stopping TPN

SUMMARY:
To provide children dependent on total parenteral nutrition with Omegaven®, a fish oil-based intravenous lipid emulsion that may be less hepatotoxic than conventional, vegetable oil-based intravenous lipid emulsions, and that may therefore reduce the need for liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* The targeted population for enrollment is the cohort of patients with TPN-dependent short bowel syndrome, defined as any pediatric patient who, following abdominal surgery, has a residual small bowel length less than 25% of that predicted for gestational age or requires postoperative TPN for more than 42 days because of gastrointestinal intolerance and who has developed TPN-associated liver disease sufficient to pose a significant risk for progression to liver failure based on the following criteria:

  * Total serum bilirubin concentration greater than 3 mg/dL after a total duration of TPN greater than 2 months in the absence of a proven episode of bacteremia within the preceding 3 weeks.

PLUS EITHER:

• Platelet count less than 200,000/μL after a total duration of TPN greater than 2 months in the absence of a proven episode of bacteremia within the preceding 3 weeks.

OR

• Serum albumin concentration less than 3.2 mg/dL after a total duration of TPN greater than 2 months in the absence of a proven episode of bacteremia within the preceding 3 weeks.

Patients with coagulopathy due to parenteral nutrition-associated liver disease (INR > 1.2) will be potential candidates for enrollment, because patients with an elevated INR exceeding 2 have demonstrated resolution of coagulopathy after treatment with Omegaven®. Similarly, patients with hyperlipidemia will be potential candidates for enrollment.

Alternatively, patients currently receiving Omegaven that was initiated at another center because of intestinal failure with liver disease that do not need to meet the lab criteria listed above. The subject may continue Omegaven under this protocol at the discretion of the Principle Investigator.

Exclusion Criteria:

Patients with a history of the following will be excluded from enrollment in this protocol:

* Allergy to fish or egg protein.
* Liver disease proven or suspected to be caused by a process other than TPN-dependent short bowel syndrome, including but not limited to hepatitis C, hepatitis B, cystic fibrosis, biliary atresia, Alagille syndrome, familial intrahepatic cholestasis, and alpha-1-antitrypsin deficiency.
* Refusal of third party providers to reimburse hospital for the cost of Omegaven®.

Ages: 2 Months to 18 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MedStar Georgetown Transplant Institute, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia